CLINICAL TRIAL: NCT04694014
Title: Emotional Intelligence Skills Leaders and Managers Need to Engage Frontline Healthcare Professionals During Covid-19 Pandemic
Brief Title: Emotional Intelligence Skills Health Leaders Need During Covid-19
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: African Wood Inc (Other)
Collaborators: Alupe University College (Unknown)
Responsible Party: Sponsor
Other Study IDs: IREC/2020/143 AN0003667W500G
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Emotional Intelligence; Leadership; Health Personnel Attitude; Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Emotional Intelligence Skills study among frontline HCW managing Covid19 in Busia Kenya: Researchers from Alupe University College will select study participants as follows 6 Clinical officers, 2 nurses, 1 nutritionist, 1 lab technician, 2 lab technologists, 7 members on the sub county surveillance Matayos, Teso north and Bunyala 2 from UHC office
  Interventions: Behavioral: EI Open ended Pre-Survey and Semi Structured Interview; Behavioral: Behavioral and Cognitive Assessment; Behavioral: Geneva Emotional Competence Test (GECO)

INTERVENTIONS:
Behavioral: EI Open ended Pre-Survey and Semi Structured Interview — Provide Interview questions via online survey with informed consent to the participants then contact a 60 minute member checking interview in person or virtually via recorded Zoom sessions for each participant
Behavioral: Behavioral and Cognitive Assessment — Use Predictive index for both cognitive and behavioral assessment of the paticipants
Behavioral: Geneva Emotional Competence Test (GECO) — Administer the Geneva Emotional Competence Test to each participant

SUMMARY:
Problem The study will address the problem that no studies have established the Emotional Intelligence (EI) skills required by leaders and managers to engage frontline healthcare professionals in crisis situation like Covid19 in Kenya Purpose The purpose of the qualitative exploratory study is to identify the EI skills Leaders and managers need to engage Frontline Healthcare Professionals in Crisis.

The Research Question is:

What are the EI skills leaders and managers need to engage frontline healthcare professionals (FHP) during crisis situations such as the Covid19 pandemic?

DETAILED DESCRIPTION:
Hypothesis The Study hypothesis that Leaders and managers with appropriate emotional intelligence skills will engage frontline healthcare professionals in crisis situations resulting in desired outcomes Data Collection The data collection will start with a primer survey on surveymonkey.com, behavioral and cognitive assessments through The Predictive Index, emotional intelligence competence assessments through emco4.com, followed by semi-structured face to face or virtual interviews with the participants. The Survey data, Assessments and the transcribed semi-structured interviews will be depersonalized and made available for subsequent researchers. The Videos if any will be destroyed three years after transcription.

Participants The 20 Participants will be selected from the population. The Study population is the number of experienced frontline healthcare professionals working in Busia County of Kenya. The County Department of Health will help in recruiting participants from doctors, nurses, and other frontline healthcare professionals.

Data Analysis The Data will be analyzed using DiscoverText.com cloud-based platform applying two rounds of coding: first in Vivo coding will be applied then prior codes will be enforced. The Vivo codes will be in the participant's word and voice. Eight priori codes will be adopted from EI literature.

Societal Benefits Society needs healthcare professionals to deal with crisis situations that place them in imperilment. The leaders have constraints of resources, time and advanced knowledge. This study seeks to seek out EI skills that will enable leaders to engage healthcare professionals while recognizing the humanity in them.

ELIGIBILITY:
Inclusion Criteria:

Experience frontline healthcare professionals working in Busia County of Kenya

Exclusion Criteria:

* None healthcare professionals
* healthcare professionals not working in Busia county

Ages: 25 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Experienced healthcare professionals practicing in Busia County Kenya. Their experience, knowledge, and insights in the interface between leaders and frontline healthcare workers will be very helpful to society at large. The 20 Participants will be selected from the population. The Study population is the number of experienced frontline healthcare professionals working in Busia County of Kenya. The County Department of Health will help in recruiting participants from doctors, nurses, and other frontline healthcare professionals
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Emotional Intelligence Competences Frontline Healthcare Professional need in their Leaders | through study completion, an average of 1 year
  The EI Competences that the participants stated that are needed from their leaders by questioner

SECONDARY OUTCOMES:
EI Competence of Participants | through study completion, an average of 1 year
  The Geneva Emotional Competence (GECO) test measure of EI for each participant compared the stated EI needed by Leaders
Participant Behavioral Analysis | through study completion, an average of 1 year
  Behavioral Outcome by Predictive Index Proprietary scale

CONTACTS AND LOCATIONS:
Overall Officials: Fabian Esamai, PhD, Principal Investigator — Alupe University College; William Okedi, PhD, Principal Investigator — Alupe University College; David F AMAKOBE, DBA, Study Director — W500G Inc - Contract Research Organization
Locations (1):
- Alupe University College, Busia, Kenya

IPD SHARING:
Plan to Share IPD: Yes
The data collection will start with a primer survey on surveymonkey.com, behavioral and cognitive assessments through The Predictive Index, emotional intelligence competence assessments through emco4.com, followed by semi-structured face to face or virtual interviews with the participants. The Survey data, Assessments and the transcribed semi-structured interviews will be depersonalized and made available for subsequent researchers. The Videos if any will be destroyed three years after transcription.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The Study report will be published six months after the end of the study. The Behavioral Assessment data, the interview results and the GECO will be depersonalized and made available on request from W500G Inc
Access Criteria: On specific request and agreement to data safety and participant privacy

REFERENCES:
- [Background] Boyatzis RE. The Behavioral Level of Emotional Intelligence and Its Measurement. Front Psychol. 2018 Aug 13;9:1438. doi: 10.3389/fpsyg.2018.01438. eCollection 2018. PMID 30150958
- [Background] Roth G, Vansteenkiste M, Ryan RM. Integrative emotion regulation: Process and development from a self-determination theory perspective. Dev Psychopathol. 2019 Aug;31(3):945-956. doi: 10.1017/S0954579419000403. Epub 2019 May 22. PMID 31113502
- [Background] Ng JY, Ntoumanis N, Thogersen-Ntoumani C, Deci EL, Ryan RM, Duda JL, Williams GC. Self-Determination Theory Applied to Health Contexts: A Meta-Analysis. Perspect Psychol Sci. 2012 Jul;7(4):325-40. doi: 10.1177/1745691612447309. PMID 26168470
- [Background] Brackett MA, Salovey P. Measuring emotional intelligence with the Mayer-Salovery-Caruso Emotional Intelligence Test (MSCEIT). Psicothema. 2006;18 Suppl:34-41. PMID 17295955
- [Background] Schlegel K, Mortillaro M. The Geneva Emotional Competence Test (GECo): An ability measure of workplace emotional intelligence. J Appl Psychol. 2019 Apr;104(4):559-580. doi: 10.1037/apl0000365. Epub 2018 Oct 22. PMID 30346195